CLINICAL TRIAL: NCT04237337
Title: Drugs for the Treatment of Multiple Sclerosis and Risk of Cancer: a Pharmacovigilance Analysis in Vigibase
Acronym: PVSEPK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-PVSEP
Record Dates: First submitted 2020-01-07; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis; Malignant Tumor
Keywords: pharmacovigilance
MeSH Terms: conditions — Multiple Sclerosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- serious cancer ICSRs (cases)
  Interventions: Other: Exposure to MS drugs
- other serious reactions ICSRs (non-cases)
  Interventions: Other: Exposure to MS drugs

INTERVENTIONS:
Other: Exposure to MS drugs — Exposure in ICSRs to MS drugs (dichotomous, exposed/not exposed), for each individual MS drug

SUMMARY:
Even though the therapeutic panel for multiple sclerosis (MS) treatment has improved in the last 20 years, safety data especially for the second-line and innovative treatments are lacking. The association between MS and cancer has long been investigated but has led to conflicting results. No studies have reported an increased risk of cancer after long-term exposure to immuno-modulators. The present study will assess whether drugs for the treatment of MS are associated with an increased risk of cancer by analyzing the disproportionality of reports in the World Health Organization (WHO) pharmacovigilance database.

DETAILED DESCRIPTION:
A case non-case study using Vigibase®, the World Health Organization Global Individual Case Safety Reports (ICSRs) database which includesreports forwarded to the WHO Uppsala Monitoring Center by national pharmacovigilance systems from over 130 countries around the world since 1967. Information on the adverse effects reported include patient demographics and medical relevant history, drugs recorded according to the WHO Drug dictionary and adverse drug reactions coded with Medical Dictionary for Regulatory Activities (MedDRA) terms will be perform.

ELIGIBILITY:
Inclusion Criteria:

* Serious cases reported in the World Health Organization (WHO) database of individual safety case report from 2000 to September 2019
* Cancer overall reported by a term included in the Standardized MedDRA query (SMQ) "Malignant tumours"

Exclusion Criteria:

- Non serious cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with a drug for the treatment of MS
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Risk of reporting cancer overall specific cancers [ Time Frame: Reported in the World Health Organization (WHO) database of individual safety case reports from 2000 to 12/31/2019 ] performing a disproportionality analysis | 2000 to 2019
  o Risk of reporting cancer overall and for specific cancer types (including breast, lung, lymphoma, cervical, melanoma and NMSC) with a specific drug of MS (β-interferon, glatiramer acetate, fumaric acid, teriflunomide, fingolimod, natalizumab, ocrelizumab or alemtuzumab) compared with the others drugs of MS

SECONDARY OUTCOMES:
Risk of reporting cancer specific cancers [ Time Frame: Reported in the World Health Organization (WHO) database of individual safety case reports from 2000 to 12/31/2019 ] performing a disproportionality analysis | 2000 to 2019
  o Risk of reporting cancer specific cancer types with a specific drug of MS compared with all other non-MS drugs performing a disproportionality analysis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dolladille C, Chretien B, Peyro-Saint-Paul L, Alexandre J, Dejardin O, Fedrizzi S, Defer G. Association Between Disease-Modifying Therapies Prescribed to Persons with Multiple Sclerosis and Cancer: a WHO Pharmacovigilance Database Analysis. Neurotherapeutics. 2021 Jul;18(3):1657-1664. doi: 10.1007/s13311-021-01073-y. Epub 2021 Jul 6. PMID 34231126